CLINICAL TRIAL: NCT02021370
Title: A Randomized, Placebo-controlled, Double-blind, Parallel Group, Multicenter Study to Investigate the Efficacy and Safety of 5 Fixed Doses of BAY85-3934 Administered Orally in the Correction of Anemia in Pre-dialysis Subjects With Chronic Kidney Disease Not Currently Treated With Erythropoiesis-stimulating Agent in Europe and Asia Pacific
Brief Title: 15141 Fixed Dose Correction / naïve and Pre Dialysis (Europe and Asia Pacific)
Acronym: DIALOGUE 1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 15141; 2013-001193-14 (EudraCT Number)
Record Dates: First submitted 2013-12-20; First posted 2013-12-27 (Estimated); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Anemia; Renal Insufficiency, Chronic
Keywords: Anemia of CKD
MeSH Terms: conditions — Anemia; Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- BAY85-3934 (25mg OD) (Experimental): 25 mg once daily (OD) of BAY85-3934 Morning: 1 tablet BAY85-3934 25 mg and 2 tablets matching placebo Evening: 3 tablets matching placebo
  Interventions: Drug: BAY85-3934; Drug: Placebo
- BAY85-3934 (50mg OD) (Experimental): 50 mg OD of BAY85-3934 Morning: 2 tablets BAY85-3934 25 mg and 1 tablet matching placebo Evening: 3 tablets matching placebo
  Interventions: Drug: BAY85-3934; Drug: Placebo
- BAY85-3934 (75mg OD) (Experimental): 75 mg OD of BAY85-3934 Morning: 3 tablets BAY85-3934 25 mg Evening: 3 tablets matching placebo
  Interventions: Drug: BAY85-3934; Drug: Placebo
- BAY85-3934 (25mg BID) (Experimental): 25 mg twice daily (BID) of BAY85-3934 Morning and evening: 1 tablet BAY85-3934 25 mg and 2 tablets matching placebo
  Interventions: Drug: BAY85-3934; Drug: Placebo
- BAY85-3934 (50mg BID) (Experimental): 50 mg BID of BAY85-3934 Morning and evening: 2 tablets BAY85-3934 25 mg and 1 tablet matching placebo
  Interventions: Drug: BAY85-3934; Drug: Placebo
- Placebo BID (Placebo Comparator): Placebo BID Morning and evening: 3 tablets of placebo matching BAY85-3934 25 mg
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BAY85-3934 — 25mg Tablet
  Arms: BAY85-3934 (25mg BID); BAY85-3934 (25mg OD); BAY85-3934 (50mg BID); BAY85-3934 (50mg OD); BAY85-3934 (75mg OD)
Drug: Placebo — Matching placebo tablet

SUMMARY:
Anaemia is a condition in which blood has a lower than normal number of red blood cells. It can also occur if red blood cells do not contain enough haemoglobin, an oxygen carrying part of blood. Anaemia is common in patients with chronic kidney disease. Healthy kidneys produce a hormone called erythropoietin, which stimulates the bone marrow to produce the proper number of red blood cells needed to carry oxygen to vital organs. Chronic kidney disease is a general term that means that the kidneys are not functioning to their full potential. The study drug, BAY85-3934, is being evaluated as a drug to increase the body's ability to produce erythropoietin.

The purpose of this study is to find out if the study drug, a tablet taken orally, is safe and effective for the treatment of anaemia associated with chronic kidney disease.

The study will enroll 120 patients at multiple locations in Europe, Asia and Australia. Participation will involve a screening visit and between 12 and 14 study visits scheduled over a period of approximately 5 to 7 months. The estimated total duration of study treatment will be 16 weeks. During these scheduled visits patients will undergo a number of procedures to confirm efficacy and safety of the study drug, including measurement of heart rate and blood pressure, physical examination, Electrocardiogram and blood/urine sample collection for laboratory tests.

The study will be conducted at 5 hospitals in the UK. Bayer HealthCare AG is funding this research.

ELIGIBILITY:
Inclusion Criteria:

* Women without childbearing potential
* Male or female subjects ≥ 18 years of age with anemia of chronic kidney disease (CKD) at screening
* Estimated glomerular filtration rate of < 60 mL/min/1.73 m2 (Modification of Diet in Renal Disease [MDRD] or the formula according to Matsuo, et al)
* Not on dialysis and not expected to begin dialysis during the treatment period of the study (at least 16 weeks from randomization)
* Not treated with any erythropoiesis-stimulating agent (ESA) within 8 weeks before randomization
* Mean screening Hb concentration </= 10.5 g/dL
* Body weight of 45 kg to 125 kg, inclusive, at screening

Exclusion Criteria:

* Subjects with significant acute or chronic bleeding, such as overt gastrointestinal bleeding
* Chronic inflammatory disease that could impact erythropoiesis (e.g., systemic lupus erythematosis, rheumatoid arthritis, celiac disease) even if it is currently in remission
* Previous or concurrent cancer except cervical carcinoma in situ, treated basal cell carcinoma, superficial bladder tumors (Ta, Tis, and T1) or any cancer curatively treated > 3 years prior to randomization
* Subjects treated with any ESA within the 8 weeks before randomization
* Red blood cell (RBC) containing transfusion within the 8 weeks before randomization
* History of cardio- (cerebro-) vascular events (e.g., unstable angina, myocardial infarction, stroke, transient ischemic attack, deep vein thrombosis, pulmonary embolism) within the last 6 months from initial screening visit
* Severe rhythm or conduction disorders (e.g., HR < 50 or > 110 bpm, atrial flutter, prolonged QT > 500 msec, third degree atrioventricular [AV] block)
* New York Heart Association Class III or IV congestive heart failure
* Severe hepatic insufficiency (defined as alanine aminotransferase [ALT] or aspartate aminotransferase [AST] > 3 x the upper limit of normal [ULN], total bilirubin > 2 mg/dL, or Child-Pugh B and C) or active hepatitis, in the investigator's opinion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2014-02-10 (Actual); Primary Completion 2015-09-15 (Actual); Study Completion 2015-09-23 (Actual)

PRIMARY OUTCOMES:
Change in local laboratory hemoglobin level from baseline to the average during the last 4 weeks treatment period | Baseline and week 12 to 16

SECONDARY OUTCOMES:
Change in local laboratory hemoglobin level from baseline | Baseline up to 12 weeks
Speed of change in hemoglobin level per unit time | Up to 16 weeks
Duration of treatment exposure | Up to 16 weeks
Number of participants with serious adverse events as a measure of safety and tolerability | Up to 16 weeks
Pharmacodynamics characterized by erythropoietin concentration | Several time points up to 16 weeks
Pharmacodynamics characterized by reticulocyte count | Several time points up to 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (54):
- Australia (2):
  - Gosford, New South Wales
  - Melbourne, Victoria
- Bulgaria (6):
  - Gabrovo
  - Lovech
  - Montana
  - Pazardzhik
  - Stara Zagora
  - Veliko Tarnovo
- Limoges Cedex1, France
- Germany (4):
  - Villingen-Schwenningen, Baden-Wurttemberg
  - Bonn, North Rhine-Westphalia
  - Düsseldorf, North Rhine-Westphalia
  - Halle, Saxony-Anhalt
- Hungary (3):
  - Baja
  - Budapest
  - Pécs
- Israel (3):
  - Ashkelon
  - Hadera
  - Nahariya
- Italy (5):
  - Napoli, Campania
  - Modena, Emilia-Romagna
  - Cremona, Lombardy
  - Pavia, Lombardy
  - Livorno, Tuscany
- Japan (10):
  - Kitakyushu, Fukuoka
  - Ōkawa, Fukuoka
  - Muroran, Hokkaido
  - Hakusan, Ishikawa-ken
  - Morioka, Iwate
  - Kamakura, Kanagawa
  - Kuwana, Mie-ken
  - Chiba
  - Fukuoka
  - Nara
- Poland (6):
  - Bialystok
  - Malbork
  - Poznan
  - Radom
  - Szczecin
  - Żyrardów
- Romania (4):
  - Bucharest
  - Constanța
  - Oradea
  - Târgu Mureş
- South Korea (2):
  - Bucheon-si, Gyeonggido
  - Seoul
- Spain (2):
  - Santiago de Compostela, A Coruña
  - L'Hospitalet de Llobregat, Barcelona
- Turkey (Türkiye) (3):
  - Ankara Univ. Medical Faculty, Ankara
  - Baskent University Medical Faculty, Ankara
  - Sifa University Medical Faculty, Izmir
- United Kingdom (3):
  - Cambridge, Cambridgeshire
  - Doncaster, South Yorkshire
  - London

REFERENCES:
- [Derived] Natale P, Palmer SC, Jaure A, Hodson EM, Ruospo M, Cooper TE, Hahn D, Saglimbene VM, Craig JC, Strippoli GF. Hypoxia-inducible factor stabilisers for the anaemia of chronic kidney disease. Cochrane Database Syst Rev. 2022 Aug 25;8(8):CD013751. doi: 10.1002/14651858.CD013751.pub2. PMID 36005278